CLINICAL TRIAL: NCT04230525
Title: Noninvasive Evaluation of Hemodynamics by Using Body Impedance Method in Patients Undergoing Urgent and Elective Cesarian Section
Brief Title: Body Impedance Method in Patients Undergoing Urgent and Elective Cesarian Section
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Zuhal Çavuş, Principal Investigator, M.D., Gaziosmanpasa Research and Education Hospital
Other Study IDs: Zuhal1
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2020-06

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bioimpedence: Noninvasive hemodynamic changes will be observed by using whole-body impedance method urgent or elective cesarian section patients under general anesthesia.
  Interventions: Diagnostic Test: non invasive whole body bioimpedence system

INTERVENTIONS:
Diagnostic Test: non invasive whole body bioimpedence system — Noninvasive hemodynamic changes will be observed by using whole-body impedance method urgent or elective cesarian section patients under general anesthesia. The whole-body bioimpedance method will be used to monitör the hemodynamic changes non invasively. This method can evaluate such as cardiac output, cardiac index, stroke volüme, stroke index, stroke volüme variations, cardiac reserve, etc. Parameters with a completely noninvasive method by using only electrots. The device consists of a laptop, a software which calculates cardiac parameters and two electrodes. The measurement is done by the following process: one of these electrodes, which looks like ECG electrodes, is stuck to the wrist and the other one to the opposite ankle or each one to two wrists.

SUMMARY:
Independent form anesthetic methods, during C/S, considering both maternal and fetal conditions, some crucial hemodynamic changes can appear and can be claimed non invasively with the whole body bioimpedance. In this research, any kind of hemodynamic difference between this method and urgent or elective C/S case will be detected and the clinic pursuit can be developed creating an advantage in favor of both maternal and fetal conditions.

DETAILED DESCRIPTION:
Independent form anesthetic methods, during C/S, considering both maternal and fetal conditions, some crucial hemodynamic changes can appear and can be claimed non invasively with the whole body bioimpedance. In this research, any kind of hemodynamic difference between this method and urgent or elective C/S case will be detected and the clinic pursuit can be developed creating an advantage in favor of both maternal and fetal conditions. Under general anesthesia, measuring the hemodynamic changes with the method of non-invasive whole-body bioimpedance system during C/S.

Detection of in which phase of operations the potential changes densify and differences between urgent and elective conditions non invasively.

ELIGIBILITY:
Inclusion Criteria:

* Must be scheduled for elective or emergency cesarean section

Exclusion Criteria:

* History of cardiac surgery, and advanced cardiac valvular disease

Ages: 18 Years to 49 Years | Sex: Female
Age Groups: Adult
Study Population: Emergency or elective cesarean patients, which are between 18-45 years of age
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2021-06-10 (Estimated)

PRIMARY OUTCOMES:
MAP | 1, 5, 15, and 30 minutes following the induction of the anesthesia
  The difference in mean arterial pressure during the cesarean section between elective and emergency ceasreansection subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa TREH, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No